CLINICAL TRIAL: NCT05368519
Title: A Single-Center Study of Brijjit® - A Force Modulating Tissue Bridge For Skin Closure in Gender-Affirming Mastectomies
Brief Title: Brijjit® for Wound Closure in Gender Affirming Mastectomies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients were not interested in participating in the study
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00304
Record Dates: First submitted 2022-05-03; First posted 2022-05-10 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Right chest with Brijjit® FMTB (Experimental): Patients will be assigned to have their right chest closure completed via Brijjit® FMTB. While the other chest (not selected for intervention) will be closed via traditional suture-based methods and will serve as an internal control.
  Interventions: Device: Brijjit®
- Left chest with Brijjit® FMTB (Experimental): Patients will be assigned to have their left chest closure completed via Brijjit® FMTB. While the other chest (not selected for intervention) will be closed via traditional suture-based methods and will serve as an internal control.
  Interventions: Device: Brijjit®

INTERVENTIONS:
Device: Brijjit® — Brijjit® is a non-invasive device which serves as a force modulating tissues bridges (FMTB) to aid in wound healing. This device used in would closure and serves to modify the mechanical forces on a wound which are implicated in adverse outcomes including scar formation and complications like wound dehiscence. Brijjit® is a flexible device which attaches via adhesive to the tissue on either side of the wound, approximates the tissue and off-loads forces.
  Other Names: Brijjit® BP100-6

SUMMARY:
This study will evaluate the use of Brijjit® for wound closure in individuals undergoing bilateral double incision gender affirming mastectomies with a single surgeon (Rachel Bluebond-Langner, MD). The study will be a randomized prospective interventional study utilizing internal controls (one side of chest receives intervention, other serves as control). Primary endpoints will include scar appearance/quality and wound complications

DETAILED DESCRIPTION:
The hypothesis of this study is that the use of Brijjit® FMTB will result in improved scar outcomes as measured by both patient and treating physician as compared to traditional suture based wound closure methods. As mentioned, at present there is no standard of care for wound closure following double incision GAM, therefore an internal control approach will be taken with patients serving as their own controls. This will be achieved by having one side of the chest receive the of Brijjit® FMTB (intervention) in addition to suture closure of the skin, while the other side will be closed with traditional methods, a combination of sutures and steri-stripsTM (control).

ELIGIBILITY:
Inclusion Criteria:

* Patient self-identifies as Transgender or Gender Expansive
* Patient will undergo primary bilateral double incision mastectomy at NYULH
* All clinical criteria to be eligible for primary mastectomy must be met
* Ability to care for donor site and adhere to wound therapy (either solo or with care-giver assistance)
* Willingness to return for scheduled follow-up visits through 1 year post-operatively
* 18 years of age or older
* English Speaking

Exclusion Criteria:

* Individuals with previously diagnosed allergies or a history of adverse effects related to adhesives / adhesive tapes
* Individuals with a history of the following prescription medication use in the last year: Accutane, Systemic glucocorticoids and/or Local glucocorticoids or immunosuppressants (i.e. topical tacrolimus, topical clindamycin etc.) at the intervention site
* Individuals with a history of significant scarring or adverse scarring (hypertrophic scars or keloid scars)
* Individuals with pre-existing scars at the GAM wound closure site
* Individuals with a disorder known to negatively affect wound healing (i.e. autoimmune disease, connective tissue disease)
* Individuals with malnutrition
* Individuals with a BMI >30 kg/m2
* Individuals with a history of radiation therapy
* Active smokers or smokeless nicotine use
* History of Previous Mastectomy
* Patient is actively immunosuppressed i.e. AIDS (HIV+ acceptable), or Systemic immunosuppressants
* Patients unable to attend post-operative follow-ups in person
* Patients with a considerable history of medical non-compliance
* Patient will receive GAM not including double incisions (i.e. periareolar)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-04-19 (Estimated); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
Subjective scar evaluation by patient outcomes using POSAS | screening/baseline visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | week 2 visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | week 4 visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | week 6 visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | week 8 visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | 3-month post-surgery visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | 6-months post-surgery visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by patient outcomes using POSAS | 12-months post-surgery visit
  Patient and Observer assessment scale (POSAS) will be used to visually assess their scar appearance and complete the 10-point scale. The patient scale will include questions regarding pain, itch, thickness, color, stiffness, irregularity, and overall opinion. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | screening/baseline visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | week 2 visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | week 4 visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | week 6 visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | week 8 visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | 3-month post-surgery visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | 6-months post-surgery visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Subjective scar evaluation by surgeon outcomes using POSAS | 12-months post-surgery visit
  Clinician will visually assess the scar appearance during the visit and complete the 10-point scale. The observer scale will include items with subcategories related to vascularity, pigmentation, relief/texture, thickness, pliability, surface area and overall opinion.Scores are tabulated out of 70. Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60.
Photographic assessment for objective scar evaluation | screening/baseline visir
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | week 2 visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | week 4 visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | week 6 visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | week 8 visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | 3-month post-surgery visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | 6-months post-surgery visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Photographic assessment for objective scar evaluation | 12-months post-surgery visit
  Standard and close-up photography (part of standard of care) will be utilized for evaluation of the appearance surgical scars. These photographs will be taken utilizing the Nikon D7200 at screening/baseline, week 2, week 4, week 6, week 8, 3-month post-surgery, 6-months post-surgery and 12-months post-surgery. There will be no statistical analyses employed on the photographs
Colorimetry of Scar | screening/baseline visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | week 2 visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | week 4 visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | week 6 visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | week 8 visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | 3-month post-surgery visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | 6-months post-surgery visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.
Colorimetry of Scar | 12-months post-surgery visit
  The Pantone SkinTone Guide is a handheld tool consisting of 110 color swatches that realistically mimic human skin tones, with stepwise variations in lightness and undertone. The guide was specifically formulated to be the closest physical representation of skin colors and is the only internationally available color standard to accurately match skin tones. Each SkinTone number is comprised of a four-digit alphanumeric number; the first two numbers reflect the hue or undertone of the skin while the second two represent the tone or lightness and darkness of the skin. This tool will be utilized to establish a clinically acceptable objective assessment for assessing the coloring of patients' scars.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Bluebond-Langner, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Thomas.Calahan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.